CLINICAL TRIAL: NCT00830596
Title: Effect of Spinal Manipulation on Sensorimotor Functions in Back Pain Patients
Acronym: D2P3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2P3; U19AT004137 (NIH)
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HVLA-SM (Active Comparator): High velocity, low amplitude lumbo-pelvic manipulation
  Interventions: Other: HVLA-SM
- LVVA-SM (Active Comparator): Low velocity, variable amplitude lumbo-pelvic manipulation
  Interventions: Other: LVVA-SM
- Sham Intervention (Placebo Comparator): Light effleurage and a sham mechanically-assisted chiropractic treatment for 2 weeks followed by full spine manipulation for 4 weeks
  Interventions: Other: Sham Intervention

INTERVENTIONS:
Other: HVLA-SM — High velocity, low amplitude lumbo-pelvic manipulation
  Arms: HVLA-SM
Other: LVVA-SM — Low velocity, variable amplitude lumbo-pelvic manipulation
  Arms: LVVA-SM
Other: Sham Intervention — 2 weeks of light effleurage and a sham mechanically-assisted chiropractic treatment followed by 4 weeks active care with full spine spinal manipulation
  Other Names: light effleurage followed by SMT
  Arms: Sham Intervention

SUMMARY:
The long-term goal for this study is to understand the physiological mechanisms of various forms of spinal manipulation in order to refine and improve this therapy for appropriately selected patients. The objective of this study is to assess the effects of high-velocity low-amplitude spinal manipulation and low-velocity variable amplitude spinal manipulation on three types of sensorimotor abilities in patients with low back pain.

DETAILED DESCRIPTION:
In collaboration with the University of Iowa, the Palmer Center for Chiropractic Research will pursue the following specific aim: To determine the effects of 2 weeks (4 applications @ 2 per week) of HVLA-SM and LVVA-SM to the lumbo-pelvic region, compared to a control group receiving light effleurage and a sham mechanically assisted adjustment, on sensorimotor function as measured by: lumbo-pelvic repositioning ability, standing postural sway and response to sudden trunk loading;

ELIGIBILITY:
Inclusion Criteria:

* 21 to 65 years old
* Low back pain (LBP) score an 11 point numerical rating scale: (must be > 4 at the Phone Screening OR Baseline 1 Visit) AND (must be > 2 at the Phone Screen, Baseline 1 AND Baseline 2 Visits)
* Acute (less than 7 days), sub-acute (7 days to 7 weeks), or chronic (more than 7 weeks) LBP matching classifications 1, 2, or 3 of the Quebec Task Force (QTF) Classification system - QTF 1: Pain without radiation, QTF 2: Pain + radiation to proximal extremity, QTF 3: Pain + radiation to distal extremity, QTF 7: Spinal stenosis
* Written informed consent (ICD1, ICD2 and ICD3)

Exclusion Criteria:

* Ongoing treatment for low back pain by other health care providers - unwillingness to postpone use of all other types of manual treatment for LBP except those provided in the study (including chiropractic and osteopathic SM, physical therapy and massage) for the duration of the study period.
* Co-morbidities Bleeding Disorders Bone and Joint Pathology Cauda Equina Syndrome Contra-indication to spinal manipulation, in general Current or Pending Litigation General Poor Health Inflammatory or Destructive tissue changes to the spine Neuromuscular Diseases Obesity Osteoporosis Peripheral Neuropathies Spinal Surgery Suspicion of drug or alcohol abuse Uncontrolled hypertension Vascular claudication
* Quebec Task Force (QTF) on Spinal Disorders QTF 4: Pain + radiation to upper/lower limb with neurologic signs QTF 5: Presumptive compression of a spinal nerve root on a simple roentgenogram QTF 6: Compression of a spinal nerve root confirmed by specific imaging techniques QTF 8: Postsurgical status, 1-6 months after intervention QTF 9: Postsurgical status, >6 months after intervention 9.1: Asymptomatic 9.2: Symptomatic QTF 10: Chronic pain syndrome QTF 11: Other diagnoses
* Pregnant or nursing women
* Pacemaker
* Inability to read or verbally comprehend English
* Any Joint Replacement
* Use of spinal manipulation within the past 4 weeks. If participants are willing to delay study enrollment until four weeks post spinal manipulative therapy, then we will schedule accordingly until this criterion is met
* Sensitivity to tape used during the biomechanical assessments
* If the Study Clinician believes that diagnostic procedures other than x-rays or dipstick urinalysis are necessary to diagnose a participant's condition, then the participant will be excluded
* Beck Depression Inventory-II greater than or equal to 29
* Retention of legal advice and an open or pending case for a health-related condition

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2007-07; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Goertz, DC, PhD, Principal Investigator — Palmer College of Chiropractic
Locations (1):
- Palmer College of Chiropractic, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the resulting manuscripts have been published, data sets will be provided for public access. Potential investigators can contact one of the Co-PIs to present their hypothesis, study design, instruments and/or data on which to focus, and resources required. Depending upon the needs and desires of the requesting party, the data that are shared may include analytic tables or de-identified or limited data sets that are transmitted to the requesting parties for additional analyses.

REFERENCES:
- [Background] Wilder DG, Vining RD, Pohlman KA, Meeker WC, Xia T, Devocht JW, Gudavalli RM, Long CR, Owens EF, Goertz CM. Effect of spinal manipulation on sensorimotor functions in back pain patients: study protocol for a randomised controlled trial. Trials. 2011 Jun 28;12:161. doi: 10.1186/1745-6215-12-161. PMID 21708042
- [Background] Vining RD, Salsbury SA, Pohlman KA. Eligibility determination for clinical trials: development of a case review process at a chiropractic research center. Trials. 2014 Oct 24;15:406. doi: 10.1186/1745-6215-15-406. PMID 25344427
- [Background] Vining R, Potocki E, Seidman M, Morgenthal AP. An evidence-based diagnostic classification system for low back pain. J Can Chiropr Assoc. 2013 Sep;57(3):189-204. PMID 23997245
- [Result] Goertz CM, Xia T, Long CR, Vining RD, Pohlman KA, DeVocht JW, Gudavalli MR, Owens EF Jr, Meeker WC, Wilder DG. Effects of spinal manipulation on sensorimotor function in low back pain patients--A randomised controlled trial. Man Ther. 2016 Feb;21:183-90. doi: 10.1016/j.math.2015.08.001. Epub 2015 Aug 8. PMID 26319101
- [Result] Vining RD, Potocki E, McLean I, Seidman M, Morgenthal AP, Boysen J, Goertz C. Prevalence of radiographic findings in individuals with chronic low back pain screened for a randomized controlled trial: secondary analysis and clinical implications. J Manipulative Physiol Ther. 2014 Nov-Dec;37(9):678-87. doi: 10.1016/j.jmpt.2014.10.003. Epub 2014 Nov 1. PMID 25455834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with acute, subacute, or chronic low back pain were recruited from local communities.
Groups:
- Sham Intervention: Light effleurage and a sham mechanically-assisted chiropractic treatment for 2 weeks followed by full spine manipulation for 4 weeks
  light effleurage followed by SMT: 2 weeks of light effleurage and a sham mechanically-assisted chiropractic treatment followed by 4 weeks active care with full spine spinal manipulation
Period: Overall Study
Arm/Group | HVLA-SM | LVVA-SM | Sham Intervention
Started | 74 | 74 | 73
Completed | 72 | 72 | 67
Not Completed | 2 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HVLA-SM | LVVA-SM | Sham Intervention | Total
Number analyzed (Participants) | 74 | 74 | 73 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (10.6) | 44.5 (10.2) | 44.4 (10.5) | 44.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 33 | 101
  Male | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Postural Sway
Description: Changes in sensorimotor function, as measured by postural sway in patients with LBP from baseline to 2 weeks. The adjusted within-group mean changes from baseline to two week follow-up are detailed below for:
  Postural sway (AP=mean excursion in the anterior-posterior direction, ML= mean excursion in the medial-to-lateral direction.
Time Frame: Baseline and 2 weeks
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | HVLA-SM | LVVA-SM | Sham Intervention
Number analyzed (Participants) | 74 | 74 | 73
mm
  Postural Sway_AP excursion - Hard (mm) | -.13 [-0.60 to 0.35] | -0.26 [-0.75 to 0.22] | -0.18 [-0.66 to 0.30]
  Postural Sway_ML excursion - Hard (mm) | -0.06 [-0.25 to 0.14] | -0.06 [-0.26 to 0.14] | -0.11 [-0.31 to 0.09]
  Postural Sway_AP excursion - Soft (mm) | -0.03 [-0.63 to 0.56] | 0.02 [-0.58 to 0.63] | -0.26 [-0.87 to 0.34]
  Postural Sway_ML excursion - Soft (mm) | 0.53 [0.09 to 0.98] | 0.51 [0.06 to 0.96] | 0.2 [-0.25 to 0.64]

2. Primary Outcome: Postural Sway Speed
Description: Changes in sensorimotor function, as measured by postural sway speed in patients with LBP from baseline to 2 weeks. The adjusted within-group mean changes from baseline to two week follow-up are detailed below for:
  Sway Speed=overall center of pressure traveling distance divided by time.
Time Frame: Baseline and 2 weeks
Measure: Mean (95% Confidence Interval); unit: mm/s
Arm/Group | HVLA-SM | LVVA-SM | Sham Intervention
Number analyzed (Participants) | 74 | 74 | 73
mm/s
  Postural Sway_ Sway speed - Hard (mm/s) | 0.02 [-1.14 to 1.18] | -0.11 [-1.29 to 1.07] | -0.23 [-1.40 to 0.94]
  Postural Sway_Sway speed - Soft (mm/s) | -0.40 [-2.53 to 1.74] | -1.71 [-3.87 to 0.46] | -0.94 [-3.10 to 1.21]

3. Primary Outcome: Response to Sudden Load, Anterior Movement in Center of Pressure Excursion in SL
Description: Changes in sensorimotor function, as measured by response to sudden load in patients with LBP from baseline to 2 weeks. The adjusted within-group mean changes from baseline to two week follow-up are detailed below for Response to sudden load [RTSL], ant. COP=anterior movement in center of pressure
Time Frame: Baseline and 2 weeks
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | HVLA-SM | LVVA-SM | Sham Intervention
Number analyzed (Participants) | 74 | 74 | 73
mm | -4.7 [-7.9 to 1.5] | -4.1 [-7.4 to 0.7] | -5.8 [-9.2 to -2.4]

4. Primary Outcome: Response to Sudden Load, Peak Muscle Response Per Side
Description: Changes in sensorimotor function, as measured by response to sudden load in patients with LBP from baseline to 2 weeks. The adjusted within-group mean changes from baseline to two week follow-up are detailed below for for Response to sudden load [RTSL] (ant. COP=anterior movement in center of pressure, L=left side of erector spinae, R=right side of erector spinae)
Time Frame: Baseline and 2 weeks
Measure: Mean (95% Confidence Interval); unit: % muscle response
Arm/Group | HVLA-SM | LVVA-SM | Sham Intervention
Number analyzed (Participants) | 74 | 74 | 73
% muscle response
  RTSL_Norm. peak muscle response - L (%) | -11.4 [-21.7 to -1.2] | 5.2 [-5.0 to 15.4] | 0.1 [-10.0 to 10.2]
  RTSL_Norm. peak muscle response - R (%) | 3.4 [-3.0 to 9.8] | 1.4 [-5.2 to 8.0] | -1.2 [-7.8 to 5.3]

5. Primary Outcome: Response to Sudden Load Response Times
Description: as for outcome 4
Time Frame: Baseline and 2 weeks
Measure: Mean (95% Confidence Interval); unit: ms
Arm/Group | HVLA-SM | LVVA-SM | Sham Intervention
Number analyzed (Participants) | 74 | 74 | 73
ms
  RTSL_Response start time - L (ms) | -18.3 [-54.2 to 17.7] | -42.8 [-82.4 to -3.2] | -19.8 [-53.0 to 13.3]
  RTSL_Response start time R (ms) | -5.9 [-25.1 to 13.2] | -17.1 [-38.4 to 4.3] | -20.8 [-38.9 to -2.7]
  RTSL_Peak response time - L (ms) | -14.6 [-49.6 to 20.3] | -25.2 [-63.7 to 13.3] | -28.5 [-60.7 to 3.7]
  RTSL_Peak response time - R (ms) | -18.1 [-30.5 to -5.8] | -2.2 [-15.9 to 11.6] | 1.9 [-9.9 to 13.8]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Any untoward medical occurrence that may present itself during the conduct of the study which may or may not have a causal relationship with the study procedures.
  *The total number of AEs may exceed the total # of people affected because some people experienced multiple AEs.
Groups:
- HVLA-SM*: High velocity, low amplitude lumbo-pelvic manipulation
  HVLA-SM: High velocity, low amplitude lumbo-pelvic manipulation
- LVVA-SM*: Low velocity, variable amplitude lumbo-pelvic manipulation
  LVVA-SM: Low velocity, variable amplitude lumbo-pelvic manipulation
- Sham Intervention*: Light effleurage and a sham mechanically-assisted chiropractic treatment for 2 weeks followed by full spine manipulation for 4 weeks
  light effleurage followed by SMT: 2 weeks of light effleurage and a sham mechanically-assisted chiropractic treatment followed by 4 weeks active care with full spine spinal manipulation
Arm/Group | HVLA-SM* | LVVA-SM* | Sham Intervention*
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74 | 0/73
Other Adverse Events (participants affected / at risk) | 50/74 | 57/74 | 46/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HVLA-SM* (N=74) | LVVA-SM* (N=74) | Sham Intervention* (N=73)
Spine-related pain (Musculoskeletal and connective tissue disorders) | 46 (92) | 54 (124) | 38 (70)
Spine-related pain with radiation (Musculoskeletal and connective tissue disorders) | 8 (9) | 15 (20) | 15 (17)
Extremity pain (Musculoskeletal and connective tissue disorders) | 13 (17) | 13 (24) | 13 (18)
Headache (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 4 (5)
General stiffness/tightness (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6) | 7 (10)
Transient muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle spasm/cramp (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 2 (2)
Muscle pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (2)
Tiredness/fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness/imbalance/vertigo (General disorders) | 0 (0) | 1 (1) | 3 (4)
Nausea (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion/respiratory symptoms/allergy (General disorders) | 2 (2) | 6 (6) | 2 (2)
Migraine (General disorders) | 0 (0) | 0 (0) | 1 (1)
Insect bite (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth/facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Numbness/tingling (General disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes